CLINICAL TRIAL: NCT04586114
Title: Effect of Early Corticosteroid Therapy on Mortality in Patient With Acute Respiratory Distress Syndrome Secondary to Covid-19
Brief Title: Effect of Corticosteroid Treatment on Prognosis in ARDS Secondary to Covid-19
Acronym: CoCovSDRA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI109
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Acute Respiratory Distress Syndrome Secondary to Covid-19
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early corticosteroid: Corticosteroid treatment within first seven days after ICU admission
  Interventions: Drug: Corticosteroids and Derivatives
- Late corticosteroid: Corticosteroid treatment later than seventh day's after ICU admission
  Interventions: Drug: Corticosteroids and Derivatives
- No corticosteroid: No corticosteroid treatment during ICU stay

INTERVENTIONS:
Drug: Corticosteroids and Derivatives — Any systemic corticosteroid treatment administrated during ICU stay
  Groups: Early corticosteroid; Late corticosteroid

SUMMARY:
Study conducted on hospitalized patient in critical ill units in Nancy and Metz to evaluate if early corticosteroid treatment in first seven days after admission improve patients outcome in Acute Respiratory Distress Syndrome secondary to Covid-19 compared to later corticosteroid therapy or no treatment. Also comparison of acquired infection with or without corticosteroid treatment during hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* ICU hospitalized with acute respiratory distress syndrome secondary to Sars-Cov-2 infection diagnosed by PCR test
* Hospitalized from 01/03/2020 to 30/04/2020

Exclusion Criteria:

* Mechanical ventilation more than 48 hours at admission
* Transfert to another ICU during stay for bed management
* Corticosteroid treatment at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient more than 18 years old hospitalized in ICU from 01/03/2020 to 30/04/2020 with acute respiratory distress syndrome secondary to Sars-Cov-2 infection without any corticosteroid treatment before admission, excluding patients with mechanical ventilation more than 48 hours before admission and patients transferred to other ICU.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality in ICU | within ICU stay, on average 15 days
  Mortality rates in ICU in each group

SECONDARY OUTCOMES:
Mortality d28 | 28 days
  mortality at day 28 after ICU admission
acquired infections incidence | 28 days
  cumulative incidence of infection acquired during ICU stay
antibiotics duration | 28 days
  number of treatment days with antibiotics during ICU stay
mechanical ventilation duration | 28 days
  number of days of treatment by mechanical ventilation during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien GIBOT, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Hopital Central, Service de Reanimation Medicale, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided